CLINICAL TRIAL: NCT02165982
Title: Intensity and Dependence to Physical Activity and Its Links With Clinical and Emotional Statuses in Comparison With Healthy Controls.
Brief Title: Characteristics of Intensity and Dependence to Physical Activity in Anorexia Nervosa
Acronym: HAP-AM
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-02
Record Dates: First submitted 2014-05-02; First posted 2014-06-18 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients controles: Inpatients suffering from anorexia nervosa at Institut Mutualiste Montsouris
- Individus sains témoins: Healthy controls selected from the general population

SUMMARY:
Etude d'épidémiologie clinique multicentrique (IMM), naturalistique, comparant un échantillon clinique à un échantillon de témoins issus de la population générale.

Cette recherche se fixe pour objectif principal de déterminer, sur un large échantillon de patients pris en charge pour anorexie mentale dans des unités de soins spécialisées, les caractéristiques de l'activité physique et la dépendance à l'exercice physique en comparaison avec des sujets issus de la population générale appariés pour l'âge et le sexe.

Nous faisons l'hypothèse que les patients anorexiques mentaux sont plus actifs et plus dépendants à l'exercice physique que des sujets de la population générale de même âge et de même sexe.

ELIGIBILITY:
Inclusion Criteria:

* Sujets de sexe masculin et féminin, âgés entre 13 et 23 ans.
* Donnant leur consentement éclairé (et celui des parents pour les mineurs)
* Pour l'échantillon clinique : prise en charge pour Anorexie Mentale (selon les critères DSM-IV) dans le département de psychiatrie de l'enfant et de l'adolescent de l'Institut Mutualiste Montsouris.
* Pour l'échantillon témoin : Sujets issus de la population générale (collégiens lycéens étudiants).

Exclusion Criteria:

* Personnes refusant la recherche
* Personnes souffrant d'une condition médicale majeure ou d'une invalidité.

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pour l'échantillon clinique (patients témoins et contrôles) : prise en charge pour Anorexie Mentale (selon les critères DSM-IV) dans le département de psychiatrie de l'enfant et de l'adolescent de l'Institut Mutualiste Montsouris.
  Pour l'échantillon individus sains témoins : Sujets issus de la population générale (collégiens lycéens étudiants).
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
GPAQ-OMS | At initial assessment and 6 weeks later
  Questionnaire de l'OMS sur la pratique d'activités physiques
GLTEQ | At initial assessment and 6 weeks later
  Godin Leisure-Time Exercise Questionnaire
EDS-R | At initial assessment and 6 weeks later
  Exercise-Dependence Scale-Revised
EDQ | At initial assessment and 6 weeks later
  Exercise-Dependence Questionnaire ; sélection des questions sur les motivations à pratiquer
EDE-Q | At initial assessment and 6 weeks later
  Eating Disorder Examination Questionnaire
CIDI | At initial assessment
  Composite International Diagnostic Interview
MOCI | At initial assessment and 6 weeks later
  Maudsley Obsessive Compulsive Inventory

SECONDARY OUTCOMES:
HAD | At initial assessment and 6 weeks later
  Hospital Anxiety & Depression Scale
EMPF | At initial assessment and 6 weeks later
  Echelle Multidimensionnelle de Perfectionnisme de Frost
TMMS | At initial assessment and 6 weeks later
  (Trait Meta Mood Scale)
RES | At initial assessment and 6 weeks later
  (Rosenberg Self-Esteem Scale)
BSQ | At initial assessment and 6 weeks later
  (Body Shape Questionnaire)
BIA | At initial assessment and 6 weeks later
  Impedancemétrie Bioélectrique

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie GODART, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, Paris, France